CLINICAL TRIAL: NCT03078088
Title: Airway Alkalinization and Nasal Colonization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lakshmi Durairaj (Other)
Responsible Party: Sponsor-Investigator, Lakshmi Durairaj, Staff Physician, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 201608805
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Healthy Subjects; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tromethamine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- saline (Placebo Comparator): normal saline
  Interventions: Drug: Saline
- treatment (Experimental): tham
  Interventions: Drug: Tham

INTERVENTIONS:
Drug: Tham — alkalinizer
  Arms: treatment
Drug: Saline — Placebo
  Arms: saline

SUMMARY:
The study will be a randomized, cross-over study of THAM followed by saline or saline followed by THAM in human non-CF and CF subjects to assess nasal colonization

DETAILED DESCRIPTION:
16 subjects per group will be randomized to receive study drug or saline followed by a wash out period and cross-over to the other treatment, three times daily for 4 days. Nasal swab will be done at baseline and after both study treatment and saline treatment for assessment of airway colonization.

ELIGIBILITY:
Healthy subjects:

Inclusion Criteria:

* 16 subjects, aged 16-80, clinically stable with no significant changes in health status for 14 days prior to Day 1, written informed consent obtained fom subject.

Exclusion Criteria:

* Pregnant or lactating
* Use of any investigational drug and/or participated in any interventional clinical trial within 28 days prior to screening, smoked in the last 6 months.

CF subjects:

Inclusion Criteria:

* FEV1% >35%, O2 saturation >90% on room air, clinically stable with no significant changes in health status for 14 days prior to Day 1, written informed consent obtained from subject.

Exclusion Criteria:

* Same as for healthy subjects.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Nasal bacterial colonization | Day 5 of placebo or Tham intervention
  Culture

SECONDARY OUTCOMES:
Safety assessment questionnaire | Day 5 of placebo or Tham intervention
  Questionnaire for local side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of IOwa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided